CLINICAL TRIAL: NCT00001575
Title: Anti-Tac(90 Y-HAT) to Treat Hodgkin's Disease, Non-Hodgkin's Lymphoma and Lymphoid Leukemia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Thomas Waldmann, M.D., Principal Investigator, National Institutes of Health Clinical Center (CC)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 970110; 97-C-0110; NCT00019305 (obsolete NCT alias)
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Results first posted 2015-12-07 (Estimated); Last update posted 2015-12-07 (Estimated); Status verified 2015-10

CONDITIONS: Hodgkin's Disease; Lymphoma, Non-Hodgkin
Keywords: Yttrium 90; Radiolabeled; Anti -Tac; Calcium DTPA
MeSH Terms: conditions — Hodgkin Disease; Lymphoma, Non-Hodgkin | interventions — Pentetic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Anti-Tac yttrium 90-labeled humanized anti-Tac (90 Y-HAT) (Experimental): 10 mCi (if a bone marrow transplant was part of the patient's previous therapy) or 15 mCi of yttrium labeled anti-TAC; followed by calcium trisodium Inj (Ca DTPA).
  Ca-DTPA will be administered intravenously on Days 1-3 to clear the radioactive agent from the body
  Interventions: Biological: Y-90 Humanized Anti-Tac; Drug: Calcium-DTPA

INTERVENTIONS:
Biological: Y-90 Humanized Anti-Tac — 10 mCi (if a bone marrow transplant was part of the patient's previous therapy) or 15 mCi of yttrium labeled anti-TAC; followed by calcium trisodium Inj (Ca DTPA).
Drug: Calcium-DTPA — Ca-DTPA will be administered intravenously on Days 1-3 to clear the radioactive agent from the body

SUMMARY:
This study will examine the use of a radioactive monoclonal antibody called yttrium 90-labeled humanized anti-Tac (90 Y-HAT) for treating certain cancers. Monoclonal antibodies are genetically engineered proteins made in large quantities and directed against a specific target in the body. The anti-Tac antibody in this study is targeted to tumor cells and is tagged (labeled) with a radioactive substance called Yttrium-90 (Y-90). The study will determine the maximum tolerated dose of 90Y-HAT and examine its safety and effectiveness.

Patients 18 years of age and older with Hodgkin's disease, non-Hodgkin's lymphoma and lymphoid leukemia who have proteins on their cancer cells that react with anti-Tac may be eligible for this study. Candidates are screened with a medical history and physical examination, blood and urine tests, electrocardiogram (EKG), chest x-ray, computed tomography (CT) scan or ultrasound of the abdomen, positron emission tomography (PET) scan of the neck and body, and skin test for immune reactivity to antigens (similar to skin tuberculin test).

Before beginning treatment, participants may undergo additional procedures, including the following:

* Patients with suspicious skin lesions have a skin biopsy. An area of skin is numbed and a circular piece of skin about 1/4-inch diameter is removed with a cookie cutter-like instrument.
* Patients with hearing loss have a hearing test.
* Patients with neurological symptoms have a lumbar puncture (spinal tap). A local anesthetic is given and a needle is inserted in the space between the bones in the lower back where the cerebrospinal fluid circulates below the spinal cord. A small amount of fluid is collected through the needle.
* Patients who have not had a bone marrow biopsy within 6 months of screening also undergo this procedure. The skin and bone at the back of the hip are numbed with a local anesthetic and a small piece of bone is withdrawn through a needle.

Patients receive 90 Y-HAT in escalating doses to determine the highest dose that can be safely given. The first group of three patients receives a low dose and, if there are no significant side effects at that dose, the next three patients receive a higher dose. This continues with subsequent groups until the maximum study dose is reached. 90 Y-HAT is given through a vein (intravenous (IV)) over a 2-hour period. In addition, a drug called Pentetate Calcium Trisodium Inj (Ca-DTPA) is given via IV over 5 hours for 3 days to help reduce the side effects of the 90Y-HAT. In some patients, the 90 Y-HAT may also be attached to a radioactive metal called Indium-111 to monitor what happens to the injected material. During infusion of the drug, patients undergo PET scanning to trace the path of the injected material in the body. For this procedure, the patient lies in the scanner, remaining in one position during the entire infusion.

Blood and urine specimens are collected periodically over a 6-week period following the infusion to determine the level of the radioactive antibody. Bone marrow, lymph node, or skin biopsies may be done to determine how much of the antibody entered these sites. Patients whose disease remains stable or improves with therapy may receive up to six more infusions of 90 Y-HAT, with at least a 6-week interval between treatments.

DETAILED DESCRIPTION:
Background:

Cluster of differentiation 25 (CD25) is expressed on the malignant cells of patients with certain lymphoid malignancies as well as the non-malignant T cells that surround the malignant tumor cells of patients with Hodgkin's disease.

Zenapax is a humanized monoclonal antibody that binds to CD25.

Zenapax has been chemically modified by the addition of a chelating molecule to permit binding of radioactive yttrium.

The yttrium labeled Zenapax binds to CD25 to deliver radiation treatment to the tumor.

Objective:

To assess the toxicity and therapeutic efficacy of (90)Yttrium-labeled humanized anti-Tac((90)Y-HAT) in patients with Tac-expressing hematologic malignancies.

To determine the sites of localization of radiolabeled Zenapax.

Eligibility:

Patients with Hodgkin's disease and other CD25 positive lymphoid malignancies.

The patient must have a granulocyte of at least 1,200/mm^3 and a platelet count of greater than 100,000/mm^3.

Design:

Patients will be treated with 10 mCi (if a bone marrow transplant was part of the patient's previous therapy) or 15 mCi of yttrium labeled Zenapax.

Indium labeled Zenapax is given to demonstrate the antibody distribution and confirm localization at sites of tumor.

Treatment is given every six weeks if tolerated and patients will be hospitalized for about one week for each treatment.

Tumor response will be evaluated after every treatment. Stable or responding patients will continue treatment with evaluations after every cycle of treatment. Patients will be treated for up to seven cycles.

ELIGIBILITY:
* INCLUSION CRITERIA:

All patients must have a histologically confirmed diagnosis of Hodgkin's disease. Patients who have had an allogeneic or autologous transplant are eligible if they are more than 100 days post-transplant.

At least 10% of each patient's malignant cells from peripheral blood, lymph node, skin, or other extranodal sites must react with anti-Tac, as determined by immunofluorescent or immunoperoxidase staining. Because of the high incidence of Tac positivity in infiltrating T cells in Hodgkin's disease, patients with cluster of differentiation 25 (CD25) positive infiltrating T cells will be eligible even if the Hodgkin's cells are negative.

Diagnoses and Stage Disease: 1) Non-Hodgkin's Lymphoma (NHL): Patients with all histopathologic subtypes of Tac-expressing NHL are eligible. Patients with indolent NHL Stages II through IV are eligible if they have failed at least one standard therapy and have disease requiring treatment. Patients with aggressive NHL are eligible if they have relapse after standard chemotherapy and either are not eligible for or have refused salvage chemotherapy or bone marrow transplantation.

2) Hodgkin's disease: Patients who are considered to have a low potential for cure with conventional chemotherapy or radiation therapy are eligible. Specifically, patients with stages II-IV Hodgkin's disease are eligible if they have relapsed or failed to attain a complete remission after first-line chemotherapy and either are not eligible for or have refused salvage chemotherapy or bone marrow transplantation.

3) Cutaneous T-cell Lymphoma (CTCL): Patients with all stages of Tac-expressing CTCL are eligible with the exception of Stage Ia. Patients with Stages Ib through III are eligible if they have failed at least one standard therapy. Patients with stage IV are eligible regardless of whether they have had previous therapy.

4) Peripheral T-cell Lymphoma (PTCL): Patients with stages I - IV PTCL are eligible if they have relapsed after first-line chemotherapy and either are not eligible for or have refused salvage chemotherapy or bone marrow transplantation.

Other: Patients with lymphoid leukemias or lymphomas not easily classified in the above categories will be eligible providing they have failed standard therapy and are not eligible for or have refused bone marrow transplantation.

Patients must have a Karnofsky performance status of at least 50.

Patients must have a creatinine of less than 2.0 mg/dl. If they patient has an abnormally elevated creatinine a creatinine clearance must be greater than 50 ml/min.

Patients must have serum glutamic oxaloacetic transaminase (SGOT) and serum glutamic pyruvic transaminase (SGPT) less than 5 times the upper limit of normal, bilirubin less than 3.0 unless this is felt to be due to the malignancy.

Patients must not have clinical cardiac failure. Patients with symptomatic pulmonary dysfunction are eligible only if it is due to the underlying malignancy.

The patient must have a granulocyte count of at least 1,200/mm^3 and a platelet count of greater than 100,000/mm^3.

Patients must be able to understand and sign informed consent.

Breast-feeding females are not eligible for the study.

Omission of cytotoxic chemotherapy or other systemic therapy of the malignancy for 3 weeks prior to entry into trial. However, patients receiving corticosteroids will not be excluded. Patients receiving corticosteroids must be on a stable dose for at least three weeks before receiving yttrium 90-labeled humanized anti-Tac (90Y-HAT) on this study.

Patients must have a life expectancy of greater than 1 month.

Patients must be at least 18 years old.

EXCLUSION CRITERIA:

Female patients of child bearing potential will be tested for pregnancy; pregnant patients will be excluded from the study.

Patients who are human immunodeficiency virus (HIV) antibody positive.

Patients with symptomatic disease that is due to malignant involvement of the central nervous system.

Patients with active second primary cancer.

Patients receiving chronic anticoagulant therapy will be excluded from the study.

Patients requiring urgent chemotherapy or radiation therapy for management of their malignancy will be excluded.

Patients with evidence of myelodysplastic syndrome or chromosomal abnormalities in their screening bone marrow evaluation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 1997-04; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas A Waldmann, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Waldmann TA, White JD, Carrasquillo JA, Reynolds JC, Paik CH, Gansow OA, Brechbiel MW, Jaffe ES, Fleisher TA, Goldman CK, Top LE, Bamford R, Zaknoen E, Roessler E, Kasten-Sportes C, England R, Litou H, Johnson JA, Jackson-White T, Manns A, Hanchard B, Junghans RP, Nelson DL. Radioimmunotherapy of interleukin-2R alpha-expressing adult T-cell leukemia with Yttrium-90-labeled anti-Tac. Blood. 1995 Dec 1;86(11):4063-75. PMID 7492762
- [Background] Hakimi J, Chizzonite R, Luke DR, Familletti PC, Bailon P, Kondas JA, Pilson RS, Lin P, Weber DV, Spence C, et al. Reduced immunogenicity and improved pharmacokinetics of humanized anti-Tac in cynomolgus monkeys. J Immunol. 1991 Aug 15;147(4):1352-9. PMID 1869828
- [Background] Pinkus GS, O'Hara CJ, Said JW. Peripheral/post-thymic T-cell lymphomas: a spectrum of disease. Clinical, pathologic, and immunologic features of 78 cases. Cancer. 1990 Feb 15;65(4):971-98. doi: 10.1002/1097-0142(19900215)65:43.0.co;2-b. PMID 2297666
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_1997-C-0110.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All ph I pts who received an initial bone marrow transplantation received an initial dose of 10mCi followed by 15mCi. At the discretion of the PI on the basis of persistent reduced hematopoietic values, a subsequent dose may have been reduced from 15mCi to 10mCi or 5mCi. All ph II pts received at least one dose of 10mCi and/or 15mCi, or 20mCi.
Period: Overall Study
Arm/Group | Anti-Tac Yttrium 90-labeled Humanized Anti-Tac (90 Y-HAT)
Started | 87
Treated | 65
Completed | 42
Not Completed | 45
Not completed — Screening failures-Ph I portion | 22
Not completed — Withdrawn/deaths | 23

BASELINE CHARACTERISTICS:
Arm/Group | Anti-Tac Yttrium 90-labeled Humanized Anti-Tac (90 Y-HAT)
Number analyzed (Participants) | 87
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 70
  >=65 years | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 36 (16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34
  Male | 53
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 81
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 15
  White | 66
  More than one race | 0
  Unknown or Not Reported | 5
Region of Enrollment [Number; unit: participants]
  United States | 87

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of 90Y-HAT
Description: Phase I portion maximum tolerated dose (MTD) is defined as the dose level below the dose at which 2 out of 2-6 patients develop DLT (if any patient develops grade IV toxicity of any type (excluding grade IV neutropenia) or grade III non-hematologic toxicity that patient may not continue on the study at the same dose level and therefore has had a dose limiting toxicity). There can be no more than 1 out of 6 patients with DLT at the MTD. The MTD will be assessed using only the results from the first cycle of therapy.
Time Frame: Patients could receive 90Y-HAT 15mCi per cycle and complete up to a maximum of 7 doses or 2 doses by the average of every 6 weeks.
Population: Phase I portion-maximum tolerated dose. Only the Hodgkin's participants was analyzed (i.e., 28).
Measure: Number; unit: mci
Arm/Group | Anti-Tac Yttrium 90-labeled Humanized Anti-Tac (90 Y-HAT)
Number analyzed (Participants) | 28
mci | 15

2. Primary Outcome: Clinical Response
Description: Clinical Response of patient is measured by the Response Evaluation Criteria in Solid Tumors (RECIST). Tumor responses were evaluated by In-HAT imaging (i.e., simultaneous with administration of therapeutic 90Y-daclizumab), Fludeoxyglucose (18F) positron-emission tomography (FDG PET) scans and computed tomography (CT) scans. Complete response is a disappearance of all measurable and evaluable disease lasting more than I month. Partial response is a reduction by ≥ 50% of leukemic cell count or ≥ 50% reduction in the size of all measurable lesions, and no increase in size of any measurable or evaluable lesion or appearance of new lesions for 1 month. Stable disease is less than partial response with no more than a 25% increase in leukemic cell count, no new lesions, or less than a 25% increase in any measurable lesion. Progressive disease is at least a 25% increase in leukemic cell count, appearance of new lesions, or an increase of 25% or greater in any measurable lesion after 2 weeks.
Time Frame: Patient would be measured with computed tomography (CT) scan, Fludeoxyglucose (18F) positron-emission tomography (FDG PET) scan in 28 days before treatment. Patient would be evaluated with In-HAT imaging at Day 1,4,5,6 and Day 7 in week 1 of each cycle.
Population: Phase II portion. Only the Hodgkin's participants was analyzed (i.e., added more Hodgkins participants to study).
Measure: Number; unit: participants
Arm/Group | Anti-Tac Yttrium 90-labeled Humanized Anti-Tac (90 Y-HAT)
Number analyzed (Participants) | 46
participants
  Complete Response | 14
  Partial Response | 9
  Stable Disease | 14
  Progressive Disease | 9

3. Secondary Outcome: Number of Participants With Adverse Events
Description: Here is the number of participants with adverse events. For a detailed list of adverse events, see the adverse event module.
Time Frame: 16 yrs 18 days
Measure: Number; unit: participants
Arm/Group | Anti-Tac Yttrium 90-labeled Humanized Anti-Tac (90 Y-HAT)
Number analyzed (Participants) | 64
participants | 57

ADVERSE EVENTS:
Arm/Group | Anti-Tac Yttrium 90-labeled Humanized Anti-Tac (90 Y-HAT)
Serious Adverse Events (participants affected / at risk) | 8/64
Other Adverse Events (participants affected / at risk) | 49/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anti-Tac Yttrium 90-labeled Humanized Anti-Tac (90 Y-HAT) (N=64)
BLOOD/BONE MARROW:: Bone marrow cellularity (Blood and lymphatic system disorders) | 1 (1)
CARDIOVASCULAR (GENERAL):: Hypotension (Cardiac disorders) | 1 (1)
HEPATIC:: Liver dysfunction/failure (clinical) (Hepatobiliary disorders) | 1 (1)
Multi-organ failure (General disorders) | 1 (1)
PULMONARY:: Pulmonary-Other (Specify, respiratory failure) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
PAIN:: Abdominal pain or cramping (Gastrointestinal disorders) | 1 (1)
PAIN:: Pain-Other (Specify, tooth pain) (General disorders) | 1 (1)
PULMONARY:: Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
PULMONARY:: Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Secondary Malignancy-Other (Specify,____) excludes metastasis from initial primary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) — MDS
Secondary Malignancy-Other (Specify,____) excludes metastasis from initial primary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — MDS/AML
Secondary Malignancy-Other (Specify,____) excludes metastasis from initial primary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — myelodysplastic syndrome
SYNDROMES:: Syndromes-Other (Specify, MDS) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anti-Tac Yttrium 90-labeled Humanized Anti-Tac (90 Y-HAT) (N=64)
ALLERGY/IMMUNOLOGY:: Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 1 (1)
ALLERGY/IMMUNOLOGY:: Allergic rhinitis (including sneezing, nasal stuffiness, postnasal drip) (Immune system disorders) | 2 (2)
ALLERGY/IMMUNOLOGY:: Allergy-Other (Specify, sinus congestion) (Immune system disorders) | 1 (1)
AUDITORY/HEARING:: Auditory/Hearing-Other (Specify, pressure in right ear) (Ear and labyrinth disorders) | 1 (1)
BLOOD/BONE MARROW:: Hemoglobin (Blood and lymphatic system disorders) | 33 (109)
BLOOD/BONE MARROW:: Leukocytes (total WBC) (Blood and lymphatic system disorders) | 32 (132)
BLOOD/BONE MARROW:: Lymphopenia (Blood and lymphatic system disorders) | 37 (142)
BLOOD/BONE MARROW:: Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 15 (64)
BLOOD/BONE MARROW:: Platelets (Blood and lymphatic system disorders) | 37 (115)
BLOOD/BONE MARROW:: Transfusion: Platelets (Blood and lymphatic system disorders) | 1 (1)
CARDIOVASCULAR (ARRHYTHMIA):: Prolonged QTc interval (QTc > 0.48 seconds) (Cardiac disorders) | 1 (1)
CARDIOVASCULAR (ARRHYTHMIA):: Sinus bradycardia (Cardiac disorders) | 1 (1)
CARDIOVASCULAR (ARRHYTHMIA):: Sinus tachycardia (Cardiac disorders) | 1 (1)
CARDIOVASCULAR (ARRHYTHMIA):: Supraventricular arrhythmias (SVT/atrial fibrillation/flutter) (Cardiac disorders) | 1 (3)
CARDIOVASCULAR (GENERAL):: Edema (Cardiac disorders) | 4 (4)
CARDIOVASCULAR (GENERAL):: Hypotension (Cardiac disorders) | 10 (15)
COAGULATION:: Partial thromboplastin time (PTT) (Blood and lymphatic system disorders) | 10 (19)
COAGULATION:: Prothrombin time (PT) (Blood and lymphatic system disorders) | 6 (12)
CONSTITUTIONAL SYMPTOMS:: Fatigue (lethargy, malaise, asthenia) (General disorders) | 8 (9)
Fever (in the absence of neutropenia, where neutropenia is defined as AGC<1.0 x 10e9/L) (General disorders) | 18 (37) — CONSTITUTIONAL SYMPTOMS
CONSTITUTIONAL SYMPTOMS:: Rigors, chills (General disorders) | 5 (6)
CONSTITUTIONAL SYMPTOMS:: Weight loss (General disorders) | 1 (1)
DERMATOLOGY/SKIN:: Dermatology/Skin-Other (Specify, eczematoid dermatitis) (Skin and subcutaneous tissue disorders) | 1 (1)
DERMATOLOGY/SKIN:: Dermatology/Skin-Other (Specify, rash; erythematous, eczematous) (Skin and subcutaneous tissue disorders) | 1 (1)
DERMATOLOGY/SKIN:: Dermatology/Skin-Other (Specify, skin lesions) (Skin and subcutaneous tissue disorders) | 1 (1)
DERMATOLOGY/SKIN:: Flushing (Skin and subcutaneous tissue disorders) | 1 (1)
DERMATOLOGY/SKIN:: Pruritus (Skin and subcutaneous tissue disorders) | 5 (5)
DERMATOLOGY/SKIN:: Rash/desquamation (Skin and subcutaneous tissue disorders) | 8 (8)
ENDOCRINE:: Hot flashes/flushes (Endocrine disorders) | 1 (1)
ENDOCRINE:: Hypothyroidism (Endocrine disorders) | 1 (1)
GASTROINTESTINAL:: Anorexia (Gastrointestinal disorders) | 4 (4)
GASTROINTESTINAL:: Constipation (Gastrointestinal disorders) | 5 (5)
GASTROINTESTINAL:: Dehydration (Gastrointestinal disorders) | 1 (1)
GASTROINTESTINAL:: Diarrhea patients without colostomy (Gastrointestinal disorders) | 4 (5)
GASTROINTESTINAL:: Dyspepsia/heartburn (Gastrointestinal disorders) | 5 (5)
GASTROINTESTINAL:: Dysphagia, esophagitis, odynophagia (painful swallowing) (Gastrointestinal disorders) | 2 (2)
GASTROINTESTINAL:: Gastrointestinal-Other (Specify, tongue discoloration) (Gastrointestinal disorders) | 1 (1)
GASTROINTESTINAL:: Mouth dryness (Gastrointestinal disorders) | 1 (1)
GASTROINTESTINAL:: Nausea (Gastrointestinal disorders) | 15 (21)
GASTROINTESTINAL:: Taste disturbance (dysgeusia) (Gastrointestinal disorders) | 1 (1)
GASTROINTESTINAL:: Vomiting (Gastrointestinal disorders) | 12 (15)
HEMORRHAGE:: Hematuria (in the absence of vaginal bleeding) (Renal and urinary disorders) | 1 (1)
HEMORRHAGE:: Rectal bleeding/hematochezia (Gastrointestinal disorders) | 1 (1)
HEPATIC:: Alkaline phosphatase (Hepatobiliary disorders) | 12 (25)
HEPATIC:: Bilirubin (Hepatobiliary disorders) | 12 (26)
HEPATIC:: Hypoalbuminemia (Hepatobiliary disorders) | 31 (76)
HEPATIC:: SGOT (AST) (serum glutamic oxaloacetic transaminase) (Hepatobiliary disorders) | 16 (33)
HEPATIC:: SGPT (ALT) (serum glutamic pyruvic transaminase) (Hepatobiliary disorders) | 16 (23)
INFECTION/FEBRILE NEUTROPENIA:: Catheter-related infection (Infections and infestations) | 1 (1)
INFECTION/FEBRILE NEUTROPENIA:: Infection without neutropenia (Infections and infestations) | 11 (17)
METABOLIC/LABORATORY:: Amylase (Metabolism and nutrition disorders) | 3 (3)
METABOLIC/LABORATORY:: Bicarbonate (Metabolism and nutrition disorders) | 1 (1)
METABOLIC/LABORATORY:: CPK (creatine phosphokinase) (Metabolism and nutrition disorders) | 6 (7)
METABOLIC/LABORATORY:: Hypercalcemia (Metabolism and nutrition disorders) | 3 (5)
METABOLIC/LABORATORY:: Hypercholesterolemia (Metabolism and nutrition disorders) | 6 (9)
METABOLIC/LABORATORY:: Hyperglycemia (Metabolism and nutrition disorders) | 12 (19)
METABOLIC/LABORATORY:: Hyperkalemia (Metabolism and nutrition disorders) | 5 (5)
METABOLIC/LABORATORY:: Hypermagnesemia (Metabolism and nutrition disorders) | 7 (11)
METABOLIC/LABORATORY:: Hypernatremia (Metabolism and nutrition disorders) | 3 (5)
METABOLIC/LABORATORY:: Hypertriglyceridemia (Metabolism and nutrition disorders) | 3 (3)
METABOLIC/LABORATORY:: Hyperuricemia (Metabolism and nutrition disorders) | 3 (4)
METABOLIC/LABORATORY:: Hypocalcemia (Metabolism and nutrition disorders) | 12 (21)
METABOLIC/LABORATORY:: Hypoglycemia (Metabolism and nutrition disorders) | 4 (4)
METABOLIC/LABORATORY:: Hypokalemia (Metabolism and nutrition disorders) | 5 (7)
METABOLIC/LABORATORY:: Hypomagnesemia (Metabolism and nutrition disorders) | 18 (31)
METABOLIC/LABORATORY:: Hyponatremia (Metabolism and nutrition disorders) | 15 (25)
METABOLIC/LABORATORY:: Hypophosphatemia (Metabolism and nutrition disorders) | 7 (16)
METABOLIC/LABORATORY:: Lipase (Metabolism and nutrition disorders) | 2 (5)
METABOLIC/LABORATORY:: Metabolic/Laboratory-Other (Specify, low zinc) (Metabolism and nutrition disorders) | 34 (58)
METABOLIC/LABORATORY:: Metabolic/Laboratory-Other (Specify, low zinc serum) (Metabolism and nutrition disorders) | 4 (7)
METABOLIC/LABORATORY:: Metabolic/Laboratory-Other (Specify, serum zinc) (Metabolism and nutrition disorders) | 1 (1)
METABOLIC/LABORATORY:: Metabolic/Laboratory-Other (Specify, zinc) (Metabolism and nutrition disorders) | 4 (11)
METABOLIC/LABORATORY:: Metabolic/Laboratory-Other (Specify, zinc, low) (Metabolism and nutrition disorders) | 1 (1)
METABOLIC/LABORATORY:: Metabolic/Laboratory-Other (Specify, zinc-serum (low)) (Metabolism and nutrition disorders) | 1 (3)
MUSCULOSKELETAL:: Musculoskeletal-Other (Specify, Akathisia) (Musculoskeletal and connective tissue disorders) | 1 (1)
MUSCULOSKELETAL:: Musculoskeletal-Other (Specify,muscle aches) (Musculoskeletal and connective tissue disorders) | 1 (1)
MUSCULOSKELETAL:: Osteonecrosis (avascular necrosis) (Musculoskeletal and connective tissue disorders) | 1 (1)
NEUROLOGY:: Dizziness/lightheadedness (Nervous system disorders) | 3 (3)
NEUROLOGY:: Insomnia (Nervous system disorders) | 3 (3)
OCULAR/VISUAL:: Ocular/Visual-Other (Specify, transient vision lost) (Eye disorders) | 1 (1)
PAIN:: Abdominal pain or cramping (Gastrointestinal disorders) | 7 (8)
PAIN:: Arthralgia (joint pain) (Musculoskeletal and connective tissue disorders) | 3 (5)
PAIN:: Bone pain (Musculoskeletal and connective tissue disorders) | 5 (6)
PAIN:: Chest pain (non-cardiac and non-pleuritic) (Musculoskeletal and connective tissue disorders) | 3 (3)
PAIN:: Headache (Nervous system disorders) | 9 (13)
PAIN:: Myalgia (muscle pain) (Musculoskeletal and connective tissue disorders) | 10 (16)
PAIN:: Pain-Other (Specify, ankle) (General disorders) | 1 (1)
PAIN:: Pain-Other (Specify, Back) (General disorders) | 1 (1)
PAIN:: Pain-Other (Specify, jaw pain/tightness) (General disorders) | 1 (1)
PAIN:: Pain-Other (Specify, pain Lt axilla surgical site) (General disorders) | 1 (1)
PAIN:: Pain-Other (Specify, pain: Back:sacral area) (General disorders) | 1 (1)
PAIN:: Pain-Other (Specify, Rt shoulder pain) (General disorders) | 1 (1)
PAIN:: Pain-Other (Specify, Rt great toe pain: ingrown toenail) (General disorders) | 1 (1)
PAIN:: Pain-Other (Specify, Rt flank) (General disorders) | 1 (1)
PAIN:: Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
PAIN:: Tumor pain (onset or exacerbation of tumor pain due to treatment) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
PULMONARY:: Cough (Respiratory, thoracic and mediastinal disorders) | 8 (8)
PULMONARY:: Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 3 (3)
PULMONARY:: Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
PULMONARY:: Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 2 (2)
PULMONARY:: Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 1 (1)
PULMONARY:: Pulmonary-Other (Specify, upper respiratory infection) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
RENAL/GENITOURINARY:: Creatinine (Renal and urinary disorders) | 4 (10)
RENAL/GENITOURINARY:: Dysuria (painful urination) (Renal and urinary disorders) | 1 (1)
RENAL/GENITOURINARY:: Hemoglobinuria (Renal and urinary disorders) | 2 (4)
RENAL/GENITOURINARY:: Proteinuria (Renal and urinary disorders) | 1 (2)
RENAL/GENITOURINARY:: Renal/Genitourinary-Other (Specify, hesitancy) (Renal and urinary disorders) | 1 (1)
SEXUAL/REPRODUCTIVE FUNCTION:: Irregular menses (change from baseline) (Reproductive system and breast disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No